CLINICAL TRIAL: NCT01972685
Title: Comparison of Transbronchial, Cryoprobe and VATS Biopsy For the Diagnosis of Interstitial Lung Disease (ILD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00044455
Record Dates: First submitted 2013-06-27; First posted 2013-10-30 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2018-11

CONDITIONS: Interstitial Lung Disease
Keywords: ILD, transbronchial, cryoprobe, VATS
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryo vs Transbronchial vs VATS biopsy (Other): Each patient will be brought to the operating room and will undergo transbronchial, cryoprobe and VATS biopsy of the lung.
  Interventions: Procedure: Cryobiopsy biopsy; Procedure: Transbronchial Biopsy; Procedure: VATS biopsy

INTERVENTIONS:
Procedure: Cryobiopsy biopsy — Cryobiopsy vs. Transbronchial vs. VATS biopsy
Procedure: Transbronchial Biopsy
Procedure: VATS biopsy

SUMMARY:
The objective of this study is to compare the sample size, architectural preservation and diagnostic yield of bronchoscopic cryo-probe transbronchial lung biopsy (C-TBBx) to bronchoscopic standard transbronchial lung biopsy (S-TBBx) and Video-Assisted Thoracoscopic Surgery (VATS) lung biopsy for the diagnosis of interstitial lung disease (ILD).

DETAILED DESCRIPTION:
This is a prospective cohort study in which 20 subjects that have suspected ILD who are undergoing non-emergent surgical biopsy will be enrolled.

Patients who have been referred to the thoracic surgery service for VATS biopsy to diagnose suspected ILD and meet basic inclusion/exclusion criteria will be approached by the study investigators and informed of the study. An informed consent will be obtained during the clinic visit with the thoracic surgeon.

At the beginning of the surgical procedure, under general anesthesia in the operating room, patients will undergo flexible bronchoscopy through the endotracheal tube and obtain 10 standard transbronchial biopsies (S-TBBx) and 5 Cryoprobe biopsies (C-TBBx) with fluoroscopic guidance. S-TBBx will be performed using standard biopsy forceps (Boston Scientific, Natick, MA) - 2.0mm diameter. C-TBBx will be performed using the cryoprobe (ERBE, Tubingen, Germany) -1.9 mm diameter, 78cm in length. This cryoprobe is routinely used in the bronchoscopy suite for other applications such as foreign body removal and local treatment of carcinoma; therefore it is a technique already employed by the interventional pulmonologists who are familiar with its use. Once the biopsies are obtained by the interventional pulmonologist, the thoracic surgeon will perform video-assisted thoracoscopic biopsy (VATS) biopsy. Following their procedure, subjects will be monitored in the post-anesthesia care unit as per standard of care. As part of their ongoing follow-up care, all subjects will be monitored for any adverse events that may have resulted from either the surgical or bronchoscopic procedure, specifically bleeding or pneumothorax.

All biopsy samples will be analyzed by a specialist in pulmonary pathology.

The number and size of all biopsies, architectural preservation of the airways/alveoli, and pathological diagnosis will be reported by the pathologist. Diagnostic yield will be calculated for each biopsy technique and compared.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides informed consent
* Subject is >18 years of age
* Subject is scheduled to undergo VATS biopsy for suspected ILD as part of their standard medical care
* A negative pregnancy test in women of child-bearing potential
* Subject is mentally capable of understanding study procedures

Exclusion Criteria:

* Study subject has any disease or condition that interferes with safe completion of the study including:

  * Platelet count < 50,000 or Coagulopathy defined as an International Normalized Ratio (INR) > 1.5 on the day of procedure, as well as discontinuation of ticagrelor or clopidogrel within 5 days of procedure.
  * Severely impaired lung function as determined with spirometry evidenced by a forced expiratory volume in 1 second (FEV1) < 0.8, or radiographically as diffuse bullous disease
  * Hemodynamic instability with systolic blood pressure <90 mmHg or heart rate > 120 beats/min, unless deemed to be stable with these values by the surgical or interventional pulmonary attending physicians
  * Hypoxemia with pulse oximetry values <88% or partial pressure of oxygen in arterial blood (PaO2) < 60 on baseline oxygen requirements
* Concurrent participation in another study involving investigational drugs or investigational medical devices
* Inability to read and understand the necessary study documents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-06; Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Comparison of biopsy technique | Day of procedure, approximately 3 hours
  The number and size of all biopsies, architectural preservation of the airways/alveoli, and pathological diagnosis will be reported by the pathologist. Diagnostic yield will be calculated for each biopsy technique and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Momen M Wahidi, MD, MBA, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Griff S, Ammenwerth W, Schonfeld N, Bauer TT, Mairinger T, Blum TG, Kollmeier J, Gruning W. Morphometrical analysis of transbronchial cryobiopsies. Diagn Pathol. 2011 Jun 16;6:53. doi: 10.1186/1746-1596-6-53. PMID 21679402
- [Background] Babiak A, Hetzel J, Krishna G, Fritz P, Moeller P, Balli T, Hetzel M. Transbronchial cryobiopsy: a new tool for lung biopsies. Respiration. 2009;78(2):203-8. doi: 10.1159/000203987. Epub 2009 Feb 21. PMID 19246874
- [Background] Krasna MJ, White CS, Aisner SC, Templeton PA, McLaughlin JS. The role of thoracoscopy in the diagnosis of interstitial lung disease. Ann Thorac Surg. 1995 Feb;59(2):348-51. doi: 10.1016/0003-4975(94)00844-w. PMID 7847948
- [Background] Deshmukh SP, Krasna MJ, McLaughlin JS. Video assisted thoracoscopic biopsy for interstitial lung disease. Int Surg. 1996 Oct-Dec;81(4):330-2. PMID 9127787
- [Background] Krasna MJ, Deshmukh S, McLaughlin JS. Complications of thoracoscopy. Ann Thorac Surg. 1996 Apr;61(4):1066-9. doi: 10.1016/0003-4975(96)00021-5. PMID 8607657
- [Background] Aktas Z, Gunay E, Hoca NT, Yilmaz A, Demirag F, Gunay S, Sipit T, Kurt EB. Endobronchial cryobiopsy or forceps biopsy for lung cancer diagnosis. Ann Thorac Med. 2010 Oct;5(4):242-6. doi: 10.4103/1817-1737.69117. PMID 20981186
- [Result] Yarmus L, Akulian J, Gilbert C, Illei P, Shah P, Merlo C, Orens J, Feller-Kopman D. Cryoprobe transbronchial lung biopsy in patients after lung transplantation: a pilot safety study. Chest. 2013 Mar;143(3):621-626. doi: 10.1378/chest.12-2290. PMID 23328889